CLINICAL TRIAL: NCT04382131
Title: Hypertonic Saline Nasal Irrigation and Gargling for Suspected or Confirmed COVID-19: Pragmatic Web-based Bayesian Adaptive Randomised Controlled Trial (ELVIS COVID-19)
Brief Title: Hypertonic Saline Nasal Irrigation and Gargling in Suspected or Confirmed COVID-19 (ELVIS COVID-19)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC20042
Record Dates: First submitted 2020-05-08; First posted 2020-05-11 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-07

CONDITIONS: Upper Respiratory Tract Infections; Virus; COVID; Virus Shedding; Virus Diseases
MeSH Terms: conditions — Respiratory Tract Infections; Virus Diseases | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: ELVIS COVID-19 is a pragmatic web-based Bayesian adaptive randomised controlled, parallel group trial of hypertonic saline nasal irrigation and gargling (HSNIG) compared to standard care in participants with clinically suspected or confirmed COVID-19 being managed at home. Participants from Scotland will be self-recruiting via web based system which will randomise in a 1:1 ratio to perform HSNIG or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertonic saline nasal irrigation and gargling (Experimental): Participants in the intervention arm will be asked to perform hypertonic saline nasal irrigation and gargling up to 12 times daily for a maximum of 14 days or until they report that they feel well.
  Interventions: Other: NaCl Solution
- Standard Care (No Intervention): Participants in the control arm will be given standard NHS guidance for the management of their symptoms and household hygiene.

INTERVENTIONS:
Other: NaCl Solution — NaCl Solution prepared by participants at home using water and salt
  Arms: Hypertonic saline nasal irrigation and gargling

SUMMARY:
ELVIS COVID-19 is a pragmatic web-based Bayesian adaptive randomised controlled, parallel group trial of hypertonic saline nasal irrigation and gargling (HSNIG) compared to standard care in participants with clinically suspected or confirmed COVID-19 being managed at home.

DETAILED DESCRIPTION:
COVID-19, a recently identified disease, has spread worldwide rapidly and is now a pandemic. There is no cure for it yet. Though it causes mild to moderate illness in most people, it can cause serious illness and death, particularly in the elderly, those with chronic illness or a weakened immune system.

The ELVIS COVID-19 study is to find out if nasal washout (i.e. irrigation) and gargling with salt water (hypertonic saline) helps individuals with COVID-19 get better faster. Preliminary data from those with the common cold has found that nasal washouts and gargling with salty water may be helpful in reducing the length of the illness. This trial will help us find out if the same treatment is helpful in improving COVID-19 symptoms and preventing the spread of the disease.

After self-consenting online, participants will be randomised into one of two study groups. The control group will be given standard personal, household hygiene and social distancing advice. The intervention group will be taught using online videos how to prepare and perform hypertonic saline nasal irrigation and gargling (HSNIG) up to 12 times daily in addition to standard advice.

Participants in both the intervention and control groups will complete an online daily diary first thing in the morning, which will be sent to them via an email link. The diaries will be completed every day until the participant reports they are well or for a maximum of 14 days or participant withdrawal.This study will look for participants across Scotland, who are 18 years old or older and who are self-isolating with confirmed or suspected COVID-19, with symptoms that have developed no more than 48 hours before consent to the study. The study is conducted online and everything we ask participants to do will be done at home with items they will already have.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years)
* Those living within the UK
* Those self-isolating at home within 48 hours of the start of the illness with:

  1. Clinical symptoms suggestive of COVID-19 (i.e. those who have at least one of the following symptoms: recent onset of (i) new continuous cough and/or (ii) high temperature) and/or (iii) loss of, or change in, sense of smell or taste (anosmia) OR
  2. Those with virologically confirmed SARS-CoV-2 infection and clinical symptoms indicative of COVID-19 (as detailed in (a) above).
* Provision of informed consent

Exclusion Criteria:

* Onset of illness>48 hours
* Inability to consent
* Pregnancy
* Immunosuppression
* Inability to perform HSNIG
* Those taking part in another interventional medical trial
* Those without access to a supply of salt
* Those who have had a negative COVID-19 swab result for the present symptoms
* Those with suspected/confirmed COVID-19 in whom hospital admission is recommended
* Those who do not have access to email/internet
* Those living in a household with another person currently participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Time to resolution of symptoms as defined by the single question 'how unwell do you feel today'. | Maximum of 14 days
  Time until participant reports well

SECONDARY OUTCOMES:
Severity of all symptoms | 1-14 days or until the participant reports that they are well
  Recorded using validated Wisconsin Upper Respiratory Symptom Survey-24 (WURSS-24) questionnaire and daily diaries. The WURSS-24 questionnaire assesses the interference on daily life and severity of symptoms on a scale of 1 (not at all) to 7 (severe)
The length of time for individual symptoms to resolve | 1-14 days or until the participant reports that they are well
  Recorded using validated Wisconsin Upper Respiratory Symptom Survey-24 (WURSS-24) questionnaire and daily diaries. The WURSS-24 questionnaire assesses the interference on daily life and severity of symptoms on a scale of 1 (not at all) to 7 (severe)
Severity of individual symptoms | 1-14 days or until the participant reports that they are well
  Recorded using validated Wisconsin Upper Respiratory Symptom Survey-24 (WURSS-24) questionnaire and daily diaries. The WURSS-24 questionnaire assesses the interference on daily life and severity of symptoms on a scale of 1 (not at all) to 7 (severe)
Contacting healthcare (NHS 24, OOH, GP) | 1-14 days or until the participant reports that they are well
  Number of participants and frequency of contacts
Participants needing GP appointments | 1-14 days or until the participant reports that they are well
  Number of participants and frequency of contacts
Participants attending hospital | 1-14 days or until the participant reports that they are well
  Number of participants
Length of stay in hospital if admitted | 1-14 days or until the participant reports that they are well
  Number of days
Number of participants reporting over the counter medication use | 1-14 days or until the participant reports that they are well
  Number of participants
Reduction in transmission to household contacts | 1-14 days or until the participant reports that they are well
  Number of people within participant's household who develop symptoms
Number of participants reporting side effects of nasal irrigation | 1-14 days or until the participant reports that they are well
  Number of participants in intervention arm reporting side effects
Types and severity of side effects reported | 1-14 days or until the participant reports that they are well
  Participants asked if they have experienced common side effects or other and to rate the severity on a 7 point scale of 'Did not have this side effect' to 'severe'
Cost of over the counter medication used | 1-14 days or until the participant reports that they are well
  Estimated cost requested when participant states over the counter medication used

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Sheikh, Principal Investigator — University of Edinburgh
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided